CLINICAL TRIAL: NCT03024762
Title: Active Search for Pediatric HIV/AIDS (ASPA)
Acronym: ASPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research for Development International (Other)
Collaborators: Else Kröner Fresenius Foundation (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Dr Yumo, Habakkuk Azinyui, Dr Yumo, Habakkuk Azinyui, MD, MPH, Research for Development International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R4D0007/2015
Record Dates: First submitted 2016-12-06; First posted 2017-01-19 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Pediatric HIV Infection
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The intervention assessed is the targeted Provider-Initiated Testing and Counselling (tPITC) whereby HIV positive parents receiving HIV services in the hospital are invited to have their children of unknown HIV status tested for HIV. The control arm is the blanket Provider-Initiated Testing and Counselling (bPITC) whereby all children consulting in the hospital (and with unknown HIV status) are invited to test for HIV and this irrespective of the presenting complaint. The study is assessing in the same hospital the effectiveness of tPITC vs bPITC.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): The intervention arm involves children and adolescents with unknown HIV status, aged between 6 weeks to 19 years, born to parents living with HIV/AIDS. These children will be identified for HIV testing through their parents diagnosed with HIV or receiving HIV care in the hospital.
  Interventions: Procedure: targeted Provider-Initiated-Testing and Counseling (tPITC)
- Control arm (No Intervention): The control arm involves children and adolescents with unknown HIV status, aged between 6 weeks to 19 years; consulting in the hospital for any motive. These children will be recruited for HIV testing at the outpatient department (OPD) and this through their accompany parents/guardians. Care providers will be advised to propose HIV testing systematically to all children and adolescents showing up at the OPD irrespective of the chief complaint.

INTERVENTIONS:
Procedure: targeted Provider-Initiated-Testing and Counseling (tPITC) — The intervention arm involves children and adolescents with unknown HIV status, aged between 6 weeks to 19 years, born to parents living with HIV/AIDS. These children will be identified for HIV testing through their parents diagnosed with HIV or receiving HIV care in the hospital.
  Arms: Intervention arm

SUMMARY:
The Active Search for Pediatric HIV/AIDS (ASPA) aims at assessing the acceptability, feasibility and effectiveness of the targeted provider-initiated-testing and counseling (tPITC) in comparison with the blanket provider-initiated-testing and counseling (bPITC) among children and adolescents in Cameroon. The new knowledge generated will inform programming of more suitable strategies to identify HIV-infected children and adolescents and this will contribute to reducing the current global gap in HIV treatment among this subpopulation group.

DETAILED DESCRIPTION:
Introduction: Globally in 2014, the antiretroviral therapy (ART) coverage rate amongst children was 32% against 41% in adults, and in Cameroon this gap was even wider (10.4% % vs 28%). Identifying and linking children to care are key barriers to effective expansion of pediatric ART in resources-limited settings. To identify HIV-infected children and enroll positive cases in care, the World Health Organization (WHO) recommended in 2007, the provider-initiated-testing and counseling (PITC) strategy. The blanket PITC (bPITC), whereby all children consulting in the health facility have to be screened for HIV requires a lot of resources in terms of HIV testing kits and supplies in addition to the increased workload on the already overburden health personnel in resource-limited settings. Conversely, the targeted PITC approach (tPITC) where children born to HIV-infected parents are offered HIV testing and counseling seems more feasible and effective. The primary objective of this study is to assess the effectiveness of tPITC in comparison with bPITC in case detection of HIV-infected children and adolescents. The secondary objective is to assess the acceptability and feasibility of tPITC in comparison with bPTIC among children and adolescents in Cameroon.

Methods:

Design: The investigator will conduct in 3 health facilities a non-randomized controlled pragmatic trial comparing the effectiveness of the targeted (intervention arm) against the blanket PITC (control arm) in case finding and linkage of HIV-infected children and adolescents in HIV treatment.

Study population: For the intervention arm, the study population will be children and adolescents between 6 weeks to 19 years born to HIV-infected parents and the control arm will be children of the same age group seeking care in the hospital irrespective of the motive of consultations.

Procedure: The study will be implemented in the Limbe Regional Hospital (South West Region), the Abong-Mbang District Hospital (East Region) and the Ndop District Hospital (North West Region) in Cameroon for a period of 36 months. Prior to the conduct of the study, health facility staff will be trained in PITC implementation. Testing kits and supplies will be made available to the site. Enrolment in the 2 arms will be done simultaneously till completion of the sample size. The HIV testing and ART eligibility assessment will be done following the national guidelines.

Sample size calculation: Based on the results of the pilot of this targeted PITC, we believe that with its implementation, the yield of newly diagnosed HIV cases amongst children should at least equal the double of the yield the blanket PITC (control arm) in same health facility. Therefore, the investigators have calculated the sample size to detect the minimum effect in the intervention group equal to at least the double of the yield in the control arm. Computing the formula for sample size calculation of 2 independent samples, we obtained a sample size of 435 children per arm. Hence a total sample size of 870 children.

Data collection, management and analysis: Socio-demographic data for children and parents, HIV status and ART eligibility, linkage to care and HIV treatment outcome will be collected using standardized pre-tested questionnaires. A database will be developed on Microsoft Access for data entry. Data entry will be done progressively till the study sample size is attained. Data analysis will be done using SPSS software and findings will be reported using both descriptive and analytical statistics.

Ethical considerations: Parents' informed consent and children' assent will be required for enrollment into the study. The study will obtain an ethical clearance prior to implementation.

Outcome: This study will assess the effectiveness of targeted PITC in case identification and linkage of HIV-infected children to care/treatment. This new knowledge could be used to reduce the current global gap in pediatric and adolescent HIV treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected parents: Parents diagnosed with HIV infection or receiving HIV services in the hospital and consenting to participate will be eligible for enrollment in the study.
* Parents/guardians seeking care for their children in the hospital: Parents/guardians presenting at the hospital with sick children will be enrolled in the study irrespective of the motive of consultations for their children.
* Children of HIV infected parents: children of HIV infected parents aged between 6 weeks to 19 years old will be eligible for enrollment in the study. Parents/guardians consent will be required as well as assent of older kids.
* Children consulting in the hospital: Children aged 6 weeks to 19 years old consulting in the hospital for any reason will be eligible to participate in the study. Parents/guardians consent will be required as well as assent of older kids.
* HIV infected children: children (6weeks<years<19 years old) enrolled in HIV care in the hospital at least 2 years before the beginning of the project and after this beginning will be enrolled into the study to assess retention into care and factors associated with loss to follow up.
* Health personnel: Health personnel involved in children's consultations and consenting to participate will be enrolled in the study.

Exclusion Criteria:

* Refusal to participate: health personnel, parents/guardians, children not willing to participate will be excluded from the study
* HIV Status: Children with known HIV positive status will be excluded for HIV testing
* Age: Children below the age of 6 weeks or above 19 years will be excluded from the study
* Health conditions: parents who are critically ill or mentally unstable will be excluded from the study

Ages: 6 Weeks to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 870 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Yield | 6 months
  Proportion of newly identified HIV cases amongst all children and adolescents eligible for HIV testing 2. Prevalence: proportion of HIV cases amongst children tested

SECONDARY OUTCOMES:
Prevalence | 6 months
  Prevalence: proportion of HIV cases amongst children and adolescents tested for HIV
Linkage | 6 months
  Linkage in care: proportion of pediatric HIV cases linked to care (CD4 testing and/or enrolment on ART)
Combined effect (tPITC+bPITC) | 6 months
  Combined effect of tPITC and bPITC: Number of children tested positive and initiated on ART in the hospital during the study as compared to historical data.
Acceptability | 6 months
  HIV testing acceptance rate: proportion of parents who accepted to have their children tested for HIV. The acceptability assesses the attitude of parents/caregivers to opt in for HIV testing of their children.
feasibility | 6 months
  HIV testing uptake: proportion of children tested amongst all eligible identified through parents in HIV care (for the targeted arm) or amongst all eligible children who visited the hospital (control arm) during the enrolment period. The feasibility outcome variable assesses the capacity of the health facility to routinely test all eligible children
Retention | 24 months
  Retention in care: proportion of cases still in care 12 and 24 months after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Habakkuk Yumo, MD, MPH, Principal Investigator — Research for Development International
Locations (3):
- Cameroon (3):
  - Abong-Mbang District Hospital, Abong Mbang, East Region
  - Ndop District Hospital, Ndop, North-West Region
  - Limbe Regional Hospital, Limbe

IPD SHARING:
Plan to Share IPD: Yes
Data can be made available to other researchers through an application addressed to the sponsor (Research for Development International) and this via the Principal Investigator (Dr Yumo Habakkuk).

REFERENCES:
- [Derived] Yumo HA, Ajeh RA, Sieleunou I, Ndenkeh JN Jr, Jordan MR, Sam-Agudu NA, Kuaban C, Loescher T. Parental and child-level predictors of HIV testing uptake, seropositivity and treatment initiation among children and adolescents in Cameroon. PLoS One. 2020 Apr 13;15(4):e0230988. doi: 10.1371/journal.pone.0230988. eCollection 2020. PMID 32282808
- [Derived] Yumo HA, Kuaban C, Ajeh RA, Nji AM, Nash D, Kathryn A, Beissner M, Loescher T. Active case finding: comparison of the acceptability, feasibility and effectiveness of targeted versus blanket provider-initiated-testing and counseling of HIV among children and adolescents in Cameroon. BMC Pediatr. 2018 Sep 25;18(1):309. doi: 10.1186/s12887-018-1276-7. PMID 30253758
- See also: Research for Development International — http://www.r4dinternational.org/